CLINICAL TRIAL: NCT06774066
Title: High Volume Image Guided Injection in Mid Portion Achilles Tendinopathy
Brief Title: High Volume Injection in Mid Portion AChilles Tendinopathy
Acronym: HighIMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malta (Other)
Responsible Party: Principal Investigator, Tiziana Mifsud, PhD candidate, University of Malta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V:15062020 7806
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-01

CONDITIONS: Mid-Portion Achilles Tendinopathy
Keywords: Achilles tendinopathy; high volume saline injection; mechanical properties; free tendon

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician and the clinician assessing mechanical and morphological changes will be blinded to treatment allocation, which will reduce observer bias in the evaluation of outcomes. Additionally, ultrasonographic images will be taken and saved for offline analysis without any identification of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Progressive rehabilitation exercise group (Active Comparator): This group will receive the standard first-line treatment, which consists of education and progressive exercise-based rehabilitation tailored to the patient. The exercises will be performed once a day and the intensity and number of repetitions will be based on the patients' status. The progressive exercise program is designed to avoid exacerbating the patient's symptoms; however, some pain is permitted during the sessions following the pain monitoring model proposed by Thomee (1997) where the pain is allowed to reach a level of 5 on the Visual Analog Scale during exercises, provided that it diminishes immediately after the session. This pain should subside by the following morning and the pain and stiffness in the Achilles tendon are not permitted to increase from one day to the next.
  Interventions: Other: Progressive rehabilitation exercise programme
- High volume image guided injection + progressive rehabilitation exercise group (Experimental): The intervention group will be given the high volume image-guided injection only once at the beginning of the trial, together with the same education and progressive exercise-based rehabilitation as the control group. The participants will be informed to rest for the first three days and then start slowly the progressive exercises on the same principle as for the control group.
  Interventions: Other: High volume image guided injection; Other: Progressive rehabilitation exercise programme

INTERVENTIONS:
Other: High volume image guided injection — High volume image guided injection consists of 9.5ml of bupivacaine, 0.5ml 20mg Depo-medrol, and 40ml of injectable saline. This procedure will be commenced with a thorough disinfection of the injection site. The mid-portion of the Achilles tendon will then be imaged in the short axis to obtain a cross-sectional view of the tendon, alongside the anterior region, including Kager's fat pad, particularly in areas of maximal pain and increased neovascularity. Once the needle is correctly positioned, the high-volume fluid will be infiltrated under pressure, with ultrasound guidance confirming the reduction or complete disappearance of neovascularisation.
  Arms: High volume image guided injection + progressive rehabilitation exercise group
Other: Progressive rehabilitation exercise programme — A comprehensive explanation of the progressive exercise program will be provided to patients, along with a detailed booklet that includes four tiers of exercises, ranging from the easiest to the most challenging. Exercises include several eccentrics, isometrics and heavy slow resistance exercises. These exercises are to be performed once a day and the intensity and number of repetitions will be based on the patients' status. The progressive exercise program is designed to avoid exacerbating the patient's symptoms; however, some pain is permitted during the sessions following the pain monitoring model proposed by Thomee (1997)

SUMMARY:
This prospective randomised clinical trial aims to evaluate the effectiveness of treatment for mid-portion Achilles tendinopathy in a real-world clinical setting, minimising the excessive control typically associated with explanatory studies. The primary focus is to assess the mechanical effects of high-volume image-guided injection in combination with rehabilitation exercises over three months. Additionally, the study will determine the overall clinical improvement in participants. The main questions it aims to answer are:

Is high-volume image-guided injection treatment superior to the usual care in treating mid-portion Achilles tendinopathy? Do mechanical and morphological properties of the tendon change after the treatment?

DETAILED DESCRIPTION:
The objectives of this trial are to

* Evaluate the effectiveness of high-volume image-guided injection combined with rehabilitation exercises in improving symptoms and functionality in patients with mid-portion Achilles tendinopathy.
* Measure changes in the mechanical properties of the Achilles tendon, including dynamic stiffness, as well as morphological characteristics such as thickness, cross-sectional area, and neovascularisation following treatment.
* Assess patient-reported outcomes related to pain, disability and function using validated questionnaires
* Explore participants' experiences and perceptions regarding their symptoms and the trial itself.

ELIGIBILITY:
Inclusion Criteria:

* Participants with mid-portion Achilles tendon pain in one or both legs. In bilateral symptoms, the most symptomatic leg will be considered for assessing the intervention or standard progressive rehabilitation exercise programme.
* Participants with chronic Achilles tendinopathy for more than three months who had previously undergone physiotherapy and exercise rehabilitation but experienced no improvement or continued to suffer from severe pain.
* Having one or more ultrasonography characteristics of mid-portion tendinopathy including thickened tendon, neovascularisation, hypoechogenic areas or loss of fibrillar homogeneity.

Exclusion Criteria:

* History of previous Achilles tendon rupture or surgically repaired tendons.
* Presentation of insertional Achilles tendinopathy or concurrent pain at both the insertional and mid-portion of the Achilles tendon at the start of the study.
* Presence of neurological or metabolic conditions known to affect tendon health

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Mechanical properties of tendon - dynamic stiffness | This outcome will be measured at baseline, after 2 weeks, after 6 weeks and after 12 weeks.
  Dynamic stiffness measured using the MyotonPRO at the middle part of the free tendon and over the soleus tendinous junction as identified by ultrasonography in both short and long axis.
The Victorian Institute of Sport Assessment - Achilles | This outcome will be measured at baseline, after 2 weeks, after 6 weeks and after 12 weeks.
  The questionnaire encompasses three key domains: pain, functional capacity, and activity level, thereby providing a comprehensive assessment of the patient's condition from their perspective. The Victorian Institute of Sport Assessment - Achilles score ranges from 0 to 100, with 0 indicating no activity and maximum pain, while a score of 100 represents the highest level of activity with no pain experienced. A minimal detectable change of 12 points was considered for the change to be clinically significant (McCormack et al., 2015).

SECONDARY OUTCOMES:
Single heel raises | This outcome will be measured at baseline, after 2 weeks, after 6 weeks and after 12 weeks.
  The single-leg heel raise test was utilised to assess the strength and endurance of the plantar flexor muscles. Participants were instructed to lift their heel to the maximum possible height for up to 25 repetitions or until the onset of discomfort or pain, whichever occurred first. A metronome was used to provide auditory feedback to help maintain a consistent pace throughout the test. A successful trial of the single-leg heel raise (SLHR) was recorded if the patient was able to maintain the set pace with the metronome (60 bpm/30 repetitions per minute) and demonstrated proper plantarflexion height and alignment. The trial was considered invalid if the patient compensated by:
  * flexing the knee,
  * using a hip propulsive strategy,
  * or losing vertical displacement due to trunk flexion (Hébert-Losier et al., 2022; Hebert-Losier et al., 2017).
Ultrasonography | This outcome will be measured at baseline, after 2 weeks, after 6 weeks and after 12 weeks.
  Ultrasonography was employed to assess secondary outcome measures, including cross-sectional area, tendon length, tendon thickness, and neovascularisation.
Tampa Scale of Kinesiophobia | This outcome will be measured at baseline, after 2 weeks, after 6 weeks and after 12 weeks.
  Tampa Scale of Kinesiophobia will be used to assess patients' perspectives on their condition and the avoidance and fear of movement.
Global scale of change | This outcome will be measured after 2 weeks, after 6 weeks and after 12 weeks.
  The global rating of change consists of a single question addressing the overall change in Achilles tendon symptoms from the start of treatment to the follow-up appointment, focusing on the patient's self-perceived change in health status.

OTHER OUTCOMES:
Use of other co-interventions | This outcome will be measured after 2 weeks, after 6 weeks and after 12 weeks.
  Patients were asked to report any co-interventions undertaken during the 3-month period
Adherence to exercises | This outcome will be measured after 2 weeks, after 6 weeks and after 12 weeks.
  Participants self-reported their adherence using a 4-point Likert scale, which categorised adherence into four distinct levels: very good adherence, indicating consistent engagement with the prescribed exercise regimen; good adherence, reflecting regular participation but not on a daily basis; poor adherence, suggesting infrequent engagement; and very poor adherence, denoting minimal or no participation in the prescribed exercises. Participants were informed about the option to maintain a logbook of exercises performed; however, this was not mandatory.
Exiting interview on patient satisfaction | This outcome will be measured at the end of the trial after 12 weeks.
  An exiting satisfactory semi structured interview was conducted with willing participants to explore patients perspective on the effectiveness of their treatment and elaborate on their results.

CONTACTS AND LOCATIONS:
Overall Officials: Tiziana Mifsud, Principal Investigator — University of Malta
Locations (1):
- Mater Dei Hospital, Msida, Malta